CLINICAL TRIAL: NCT05593276
Title: The Preliminary Effects of an Internet-delivered, Layperson Facilitated Cognitive Behavioral Therapy for Depression Among Chronically Ill Older Adults: A Pilot Randomized Controlled Trial
Brief Title: The Preliminary Effects of Empower@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWD019703-HUM00212950
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorder
Keywords: Cognitive Behavioral Therapy; Older Adults; Internet-Based Intervention; Depression; Social Isolation
MeSH Terms: conditions — Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders; Social Isolation

STUDY DESIGN:
Intervention Model Description: The purpose of this research project is to assess the effectiveness of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. The program is intended to decrease depression in participants by encouraging them to participate in meaningful and enjoyable activities while challenging problematic thinking patterns.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist (No Intervention)
- Internet-based program (Experimental)
  Interventions: Behavioral: Empower@Home

INTERVENTIONS:
Behavioral: Empower@Home — Participants will be provided with access to a 9-session online program and will receive supportive remote assistance throughout regarding technical and programmatic issues.
  Arms: Internet-based program

SUMMARY:
This randomized pilot trial uses a waitlist control parallel design of a novel internet-based cognitive behavioral therapy program for older adults with elevated depressive symptoms. This study will enroll approximately 35 older adults per group throughout Michigan. The intervention will take approximately ten weeks to complete. Participants will have lower levels of depression after completing the intervention than before enrollment. Participants will be able to use the internet-based platform with minimal support.

DETAILED DESCRIPTION:
Depression affects up to 40% of homebound seniors, but most homebound seniors do not receive psychotherapy due to various access barriers. The study team focuses on developing community-based solutions to reduce these access barriers. In a previously approved project HUM00207612, the study team tested the feasibility of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. The pilot project allowed for refining study procedures and the web platform used to deliver the program. In this new project, the study team will conduct a pilot randomized control trial to test the effectiveness of Empower@Home with older adults. Recruitment methods include 1) referrals from social service agencies, 2) advertisements on social media, local news outlets, and the program website, and 3) research participant registries.

The intervention involves attending up to 9 pre-recorded online therapy sessions and receiving weekly coaching calls from trained research assistants for up to 10 weeks. Participants will engage in therapy in their private homes. Three assessments are scheduled, including a comprehensive baseline, a post-test, and a 10-week follow-up. Each assessment takes about 20-40 minutes to complete over the phone.

Between Jan and Sept 2023, about 70 subjects (35 in each group) will be recruited. Participants will be randomized into the treatment group or waitlist control. The treatment group will receive the intervention immediately, whereas the waitlist control will wait for ten weeks before starting the intervention (i.e., after the 10-week "post-test"). Therefore, this is a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years
* have at least mild depressive symptoms, based on PHQ-9 >=8
* are willing to participate

Exclusion Criteria:

* Probable cognitive impairment based on the Blessed Orientation, Memory, and Concentration scale (score >9).
* They do not speak English
* have active suicidal ideation, defined as moderate to high risk based on the 6-item Columbia-Suicide Severity Rating Scale (C-SSRS)
* Have a terminal illness or unstable physical health with a high risk of hospitalization within the next 3 months
* Have severe vision impairment that can not be corrected and with no in-home help to assist them with using a mobile device
* possible substance use disorders as assessed by the 4-item CAGE screener (>=2 on the CAGE AND have not been sober for at least one year)
* Have a self reported psychotic disorder
* Currently receiving psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Change from Baseline PHQ-9 at 10 weeks
  Change in 9 item standardized measures of depressive symptom severity. PHQ-9 score ranges from 0 to 27, with a higher score indicating more severe symptoms.
Modified Treatment Evaluation Inventory | 10 weeks
  11-item Likert scale relating to acceptability of program to participant modified for older adults and the study context. The score ranges from 11 to 55, and a higher score means higher acceptability.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder Assessment-7 (GAD-7) | Change from Baseline at 10 weeks
  Change in 7-item standardized measure for severity of anxiety symptoms. GAD-7 score ranges from 0 to 21, higher score means more severe symptoms.
Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS)-Global Health | Change from Baseline at 10 weeks
  Change in 9 item standardized measure for global health. Total score ranges from 9 to 45, higher score means better global health.
Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS)-Social Isolation | Change from Baseline at 10 weeks
  Change in 8 item standardized measure for feelings of loneliness. Total score ranges from 8 to 40, higher score means higher levels of loneliness.
Change in EQ5D-5L | Change from Baseline at 10 weeks
  Change in 5 item EQ5D-5L. Higher score indicates better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Xiang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiang X, Kayser J, Turner S, Ash S, Himle JA. Layperson-Supported, Web-Delivered Cognitive Behavioral Therapy for Depression in Older Adults: Randomized Controlled Trial. J Med Internet Res. 2024 Mar 4;26:e53001. doi: 10.2196/53001. PMID 38437013
- [Derived] Kayser J, Wang X, Wu Z, Dimoji A, Xiang X. Layperson-Facilitated Internet-Delivered Cognitive Behavioral Therapy for Homebound Older Adults With Depression: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 22;12:e44210. doi: 10.2196/44210. PMID 36811937

DOCUMENTS (1):
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT05593276/ICF_000.pdf